CLINICAL TRIAL: NCT01824498
Title: Dietary Fat, Eicosanoids and Breast Cancer Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: UMN914
Record Dates: First submitted 2013-04-01; First posted 2013-04-04 (Estimated); Results first posted 2013-09-25 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Breast Cancer
Keywords: omega-3 fatty acids; sex hormones; urinary sex hormone metabolites
MeSH Terms: conditions — Breast Neoplasms | interventions — Diet, Fat-Restricted; Diet, High-Fat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Low Fat, High Fat, Low Fat High Omega 3 (Experimental): See Intervention Description
  Interventions: Other: Low Fat diet; Other: Low Fat high n3 diet; Other: High Fat Diet
- Low Fat, Low Fat High Omega 3, High Fat (Experimental): See Intervention Description
  Interventions: Other: Low Fat diet; Other: Low Fat high n3 diet; Other: High Fat Diet
- High Fat, Low Fat, Low Fat High Omega 3 (Experimental): See Intervention Description
  Interventions: Other: Low Fat diet; Other: Low Fat high n3 diet; Other: High Fat Diet
- High Fat, Low fat High Omega 3, Low Fat (Experimental): See Intervention Description
  Interventions: Other: Low Fat diet; Other: Low Fat high n3 diet; Other: High Fat Diet
- Low Fat High Omega 3, High Fat, Low Fat (Experimental): See Intervention Description
  Interventions: Other: Low Fat diet; Other: Low Fat high n3 diet; Other: High Fat Diet
- Low Fat High Omega 3, Low Fat, High Fat (Experimental): See Intervention Description
  Interventions: Other: Low Fat diet; Other: Low Fat high n3 diet; Other: High Fat Diet

INTERVENTIONS:
Other: Low Fat diet — Low fat diet = 20% fat
Other: Low Fat high n3 diet — Low Fat high n3 diet = 20% fat + 3% n3
Other: High Fat Diet — High Fat Diet = 40% fat

SUMMARY:
The primary objective of this investigation is to determine whether diets designed to increase plasma n3 concentrations (a low fat diet, with or without n3 fatty acid enrichment), will favorably affect sex hormone distribution in women in a direction associated with reduced risk of sex hormone-mediated cancer development. Specifically, we hypothesize that an increased concentration of circulating n3 fatty acids will reduce the biochemical markers associated with increased risk for developing certain sex hormone mediated cancers such as breast cancer

DETAILED DESCRIPTION:
The guiding concept of our proposal is that both the total fat and the fatty acid composition of the diet contribute to a milieu associated with the risk for sex-hormone mediated cancers. Specifically, we hypothesize that an increased concentration of circulating n3 fatty acids will reduce the biochemical markers associated with increased risk for developing certain sex hormone mediated cancers such as breast cancer. When compared with the high fat diet, we expect n3 concentrations to increase and sex hormone levels to decrease after both low fat and low fat/n3 rich diets, with the greatest response in the low fat-n3 supplemented group. The aims of this project are: 1) to evaluate the effects of total fat and n3 fatty acid consumption on plasma and urine sex hormone concentrations in postmenopausal women, 2) to evaluate the relationship between plasma concentrations of fatty acids and plasma and urinary sex hormone concentrations, and 3) to evaluate the effects of total fat and n3 fatty acid consumption on the associations between sex hormone concentrations and urinary prostaglandin E2 and thromboxane B2 concentrations.

The primary objective of this investigation is to determine whether diets designed to increase plasma n3 concentrations (a low fat diet, with or without n3 fatty acid enrichment), will favorably affect sex hormone distribution in women in a direction associated with reduced risk of sex hormone-mediated cancer development. The primary endpoints to be evaluated include plasma and urinary sex hormone concentrations as follows:

Endpoints associates with increased risk factors for breast cancer risk: plasma estradiol (E2), estrone (E1), estrone sulfate (E1 sulfate), testosterone, androstenedione, sex hormone binding globulin (SHBG), dehydroepiandrosterone (DHEA), dehydroepiandrosterone sulfate (DHEAS), Measures of estrogen action: plasma follicle stimulating hormone (FSH), urinary estrogen metabolites.

Measures of systemic arachidonic acid-derived eicosanoids: urinary bicyclo-prostaglandin E2 (PGEa), 2,3-dinor thromboxane B2 (TXB2).

Measures reflecting influence of dietary fat and fatty acid intake: plasma phospholipid, cholesterol ester, triglyceride and free fatty acid composition.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* 45 to 70 years old,
* at least one year since their last menstrual period
* not using hormone replacement therapy,
* BMI between 19 -29
* willingness to discontinue use of over-the-counter medications with anti-prostaglandin activity such as aspirin or non-steroidal anti-inflammatory medications
* consumption of a "Typical " American diet with no unusual dietary practices such as compliance with a strict vegetarian diet
* willingness to comply with the demands of the experimental protocol.

Exclusion Criteria:

* Smoking
* Known disease process, and 3) Use of prescription medications, including hormone replacement therapy.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2004-01; Primary Completion 2008-12 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan K Raatz, PhD, RD, Principal Investigator — USDA, GFHNRC
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] McColley SP, Georgopoulos A, Young LR, Kurzer MS, Redmon JB, Raatz SK. A high-fat diet and the threonine-encoding allele (Thr54) polymorphism of fatty acid-binding protein 2 reduce plasma triglyceride-rich lipoproteins. Nutr Res. 2011 Jul;31(7):503-8. doi: 10.1016/j.nutres.2011.06.003. PMID 21840466
- [Background] Raatz SK, Young LR, Picklo MJ Sr, Sauter ER, Qin W, Kurzer MS. Total dietary fat and fatty acid content modifies plasma phospholipid fatty acids, desaturase activity indices, and urinary prostaglandin E in women. Nutr Res. 2012 Jan;32(1):1-7. doi: 10.1016/j.nutres.2011.12.006. PMID 22260857
- [Background] Young LR, Raatz SK, Thomas W, Redmon JB, Kurzer MS. Total dietary fat and omega-3 fatty acids have modest effects on urinary sex hormones in postmenopausal women. Nutr Metab (Lond). 2013 Apr 23;10(1):36. doi: 10.1186/1743-7075-10-36. PMID 23618064
- [Result] Young LR, Kurzer MS, Thomas W, Redmon JB, Raatz SK. Effect of dietary fat and omega-3 fatty acids on urinary eicosanoids and sex hormone concentrations in postmenopausal women: a randomized controlled feeding trial. Nutr Cancer. 2011;63(6):930-9. doi: 10.1080/01635581.2011.589957. Epub 2011 Jul 11. PMID 21745038

RESULTS

PARTICIPANT FLOW:
Recruitment Details: * 6
  * 137 participants screened, 66 did not meet criteria, 71 were eligible but 39 declined participation,32 screened in clinic but 2 didn't meet eligibility on further screen and 6 declined participation
Pre-assignment Details: Subjects enrolled prior to randomization (N=18)
Groups:
- Low Fat, High Fat, Low Fat High Omega 3; Low Fat, Low Fat High Omega 3, High Fat; High Fat, Low Fat, Low Fat High Omega 3; High Fat, Low Fat High Omega 3, Low Fat; Low Fat High Omega 3, High Fat, Low Fat; Low Fat High Omega 3, Low Fat, High Fat: Low Fat = 20% fat High Fat = 40% fat Low Fat, high n3 diet = 20% fat + 3% n3
Period: 1st Intervention (8 Weeks)
Arm/Group | Low Fat, High Fat, Low Fat High Omega 3 | Low Fat, Low Fat High Omega 3, High Fat | High Fat, Low Fat, Low Fat High Omega 3 | High Fat, Low Fat High Omega 3, Low Fat | Low Fat High Omega 3, High Fat, Low Fat | Low Fat High Omega 3, Low Fat, High Fat
Started | 5 | 2 | 6 | 3 | 4 | 4
Completed | 5 | 2 | 6 | 3 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (8 Weeks)
Arm/Group | Low Fat, High Fat, Low Fat High Omega 3 | Low Fat, Low Fat High Omega 3, High Fat | High Fat, Low Fat, Low Fat High Omega 3 | High Fat, Low Fat High Omega 3, Low Fat | Low Fat High Omega 3, High Fat, Low Fat | Low Fat High Omega 3, Low Fat, High Fat
Started | 5 (2 dropped out) | 2 | 6 (2 dropped out) | 3 (1 dropped out) | 4 (1 dropped out) | 4
Completed | 3 | 2 | 4 | 2 | 3 | 4
Not Completed | 2 | 0 | 2 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 2 | 1 | 1 | 0
Period: 2nd Intervention (8 Weeks)
Arm/Group | Low Fat, High Fat, Low Fat High Omega 3 | Low Fat, Low Fat High Omega 3, High Fat | High Fat, Low Fat, Low Fat High Omega 3 | High Fat, Low Fat High Omega 3, Low Fat | Low Fat High Omega 3, High Fat, Low Fat | Low Fat High Omega 3, Low Fat, High Fat
Started | 3 | 2 | 4 | 2 | 3 | 4
Completed | 3 | 2 | 4 | 2 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (8 Weeks)
Arm/Group | Low Fat, High Fat, Low Fat High Omega 3 | Low Fat, Low Fat High Omega 3, High Fat | High Fat, Low Fat, Low Fat High Omega 3 | High Fat, Low Fat High Omega 3, Low Fat | Low Fat High Omega 3, High Fat, Low Fat | Low Fat High Omega 3, Low Fat, High Fat
Started | 3 | 2 | 4 | 2 | 3 | 4
Completed | 3 | 2 | 4 | 2 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: 3rd Intervention (8 Weeks)
Arm/Group | Low Fat, High Fat, Low Fat High Omega 3 | Low Fat, Low Fat High Omega 3, High Fat | High Fat, Low Fat, Low Fat High Omega 3 | High Fat, Low Fat High Omega 3, Low Fat | Low Fat High Omega 3, High Fat, Low Fat | Low Fat High Omega 3, Low Fat, High Fat
Started | 3 | 2 | 4 | 2 | 3 | 4
Completed | 3 | 2 | 4 | 2 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Fat, High Fat, Low Fat High Omega 3 | Low Fat, Low Fat High Omega 3, High Fat | High Fat, Low Fat, Low Fat High Omega 3 | High Fat, Low Fat High Omega 3, Low Fat | Low Fat High Omega 3, High Fat, Low Fat | Low Fat High Omega 3, Low Fat, High Fat | Total
Number analyzed (Participants) | 5 | 2 | 6 | 3 | 4 | 4 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 2 | 6 | 3 | 4 | 4 | 24
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (2) | 57 (2) | 57 (2) | 57 (2) | 57 (2) | 57 (2) | 57 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 6 | 3 | 4 | 4 | 24
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 2 | 6 | 3 | 4 | 4 | 24

OUTCOME MEASURES:

1. Primary Outcome: Plasma Sex Hormone Levels
Time Frame: 8 weeks
Reporting Status: Not Posted

2. Primary Outcome: E2
Description: Estradiol
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Groups:
- High Fat Diet: Hig fat diet = 40% fat
- Low Fat, High n3 Diet: Low fat, n3 diet = 20% fat + 3% n3
Arm/Group | High Fat Diet | Low Fat Diet | Low Fat, High n3 Diet
Number analyzed (Participants) | 18 | 18 | 18
pmol/L | 52.8 (5.1) | 35.6 (5.4) | 39.8 (5.1)

ADVERSE EVENTS:
Groups:
- Low Fat, High n3 Diet: Low fat, high n3 diet = 20% fat + 3% n3
Arm/Group | High Fat Diet | Low Fat Diet | Low Fat, High n3 Diet
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No